CLINICAL TRIAL: NCT02839798
Title: Evaluation of NeoSync EEG Synchronized TMS For the Treatment of Major Depressive Episode in Bipolar Disorder and Associated Neural Response: An Open Label Trial
Brief Title: NeoSync TMS Treatment for Bipolar I Depression
Acronym: NESTTBID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding and staffing
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Linda L Carpenter MD, Chief, Mood Disorder Research Program, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1601-004
Record Dates: First submitted 2016-06-07; First posted 2016-07-21 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Major Depressive Episode; Bipolar Depression; Bipolar Disorder; Mood Disorders
Keywords: sTMS; NEST; NeoSync; synchronous; non-invasive neuromodulation; TMS; transcranial magnetic stimulation; EEG; bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Open label, unblinded treatment series, all participants receive active treatment with the investigational device (NeoSync sTMS), as adjunct to ongoing stable pharmacotherapy
Oversight: Data Monitoring Committee: No

ARMS (1):
- sTMS active (Experimental): Treatment with the NEST Device
  Interventions: Device: NEST (NeoSync EEG Synchronized TMS)

INTERVENTIONS:
Device: NEST (NeoSync EEG Synchronized TMS) — The NeoSync EEG Synchronized TMS (NEST) is an electromechanical medical device that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of Bipolar Depression.

SUMMARY:
This study is designed to evaluate the safety and preliminary efficacy of synchronized transcranial magnetic stimulation (sTMS) using the NeoSync EEG Synchronized TMS device (NEST) in subjects with Bipolar Disorder type I in a Major Depressive Episode. This is an open label study in which subjects will receive treatment 5 days per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following inclusion criteria to qualify for enrollment into the study:

1. 18 - 70 years of age;
2. DSM-5 primary diagnosis of Bipolar Disorder type 1 (with a documented past manic episode), currently in a Major Depressive Episode by diagnostic criteria elicited by structured clinical interview (SCID-5-RV);
3. MADRS score ≥ 20;
4. Duration of current episode >4 weeks
5. YMRS score ≤ 12;
6. baseline EEG of sufficient quality for quantitative analysis processing;
7. willing and able to adhere to the intensive treatment schedule and all required study visits;
8. currently on adequate dose of mood stabilizer with significant evidence base or FDA approval as antimanic or for maintenance therapy of bipolar disorder (e.g, valproic acid/divalproex, carbamazepine, lithium, aripiprazole, ziprasidone, risperidone, quetiapine, olanzapine, asenapine, haloperidol, chlorpromazine, paliperidone, cariprazine).

Exclusion Criteria: Subjects will be excluded from study participation if one of the following exclusion criteria applies:

1. unable or unwilling to give informed consent;
2. diagnosed with current primary psychotic disorder (rather than BD);
3. diagnosed with current mania or hypomanic mood episode;
4. history of moderate to severe substance use disorder within the past 6 months (except nicotine and caffeine);
5. currently being treated with a stimulant;
6. clinically defined major neurological disorder; including, but not limited to, seizure disorder and history of loss of consciousness due to head injury for greater than 10 minutes, or with documented evidence of brain injury;
7. increased risk of seizure for any reason, including diagnosis of increased intracranial pressure, comorbid neurological disorder, use of certain medications, highly unstable use of alcohol or benzodiazepines;
8. initiation of new antidepressant treatments (new medication, new device-based stimulation, or new psychotherapy) within 6 weeks prior to study baseline;
9. active suicidal intent or plan as detected on screening assessments, or in the Investigator's opinion, is likely to attempt suicide within the next six months;
10. presence of implanted cardiac pacemakers, implanted medication pumps, or intracardiac lines;
11. intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head (excluding the mouth), which cannot be safely removed;
12. clinically significant unstable medical condition;
13. if female: pregnant, not using medically acceptable means of birth control, or currently breastfeeding;
14. other condition, which in the judgment of the Investigator could prevent the subject from completion of the study;
15. for participants in the MRI study: ferromagnetic metal implant or other contraindication to imaging in a 3 Tesla MRI;
16. past treatment with TMS therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05; Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carpenter, MD, Principal Investigator — Butler Hospital, Mood Disorders Research Program, Brown Department of Psychiatry and Human Behavior
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | sTMS Active
Started | 6
Completed | 4
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | sTMS Active
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
MADRS TOTAL SCORE [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) will be performed as a baseline and endpoint assessments and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. The MADRS score ranges from 0 to 60; a score of 0-6 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
  units on a scale | 39.5 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean MADRS Total Score Change (Last Observation Carried Forward)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) will be performed as a baseline and endpoint assessments and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. The MADRS score ranges from 0 to 60; a score of 0-6 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to week 6 reported
Population: Signed consent and got at least one treatment session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | sTMS Active
Number analyzed (Participants) | 6
score on a scale | -17.8 (12.2)

2. Secondary Outcome: Mean HDRS-17 Total Score Change (Last Observation Carried Forward)
Description: The Hamilton Rating Scale for Depression (HRSD-28) will be done at baseline and endpoint assessments. The HRSD-17 score, derived from the HRSD-28, will be analyzed. The HRSD-17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline and week 6
Population: signed consent and completed at least 1 treatment session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | sTMS Active
Number analyzed (Participants) | 6
score on a scale | -7.8 (6.6)

3. Secondary Outcome: Mean IDS-SR Score Change (Last Observation Carried Forward)
Description: The Inventory of Depressive Symptomatology (IDS-SR) will be performed as a baseline and after every 5 treatments. It's a standardized self-rating scale for depressive symptom severity used in many clinical trials. IDS-SR total score ranges from 0 to 84; a score of 0-13 is generally accepted to be within the normal range (or reflect clinical remission), while a score of 26 or higher indicates at least moderate severity. Single value was average mean IDS-SR score change.
Time Frame: Baseline through week 6
Population: signed consent and completed at least 1 treatment session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | sTMS Active
Number analyzed (Participants) | 6
score on a scale | -7.7 (8.5)

ADVERSE EVENTS:
Time Frame: From Treatment Session #1 until Treatment #30 (6 weeks or LOCF if early termination)
Description: participants were queried at each treatment session
Groups:
- ACTIVE sTMS: Active Open Label Treatment with the NEST Device
  NEST (NeoSync EEG Synchronized TMS): The NeoSync EEG Synchronized TMS (NEST) is an electromechanical medical device that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of Bipolar Depression.
Arm/Group | ACTIVE sTMS
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTIVE sTMS (N=6)
dizziness or lightheadedness (Nervous system disorders) | 2 (2)
panic or anxiety attack (Nervous system disorders) | 2 (2)
headache (Nervous system disorders) | 3 (3)
Gastrointestinal upset or nausea (Gastrointestinal disorders) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Diminished Attention (Psychiatric disorders) | 1 (1)
Sinus Congestion (Ear and labyrinth disorders) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There was no external funding obtained for this trial. Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT02839798/Prot_SAP_ICF_000.pdf